CLINICAL TRIAL: NCT01577901
Title: Consumer in Stream and Container Collected Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROTOCOL-0425
Record Dates: First submitted 2012-04-11; First posted 2012-04-16 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-07

CONDITIONS: Determination of Pregnancy Status
Keywords: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Clearblue Advanced — Pregnancy test

SUMMARY:
Female volunteers, requiring to conduct a personal pregnancy test will use Clearblue Advanced Pregnancy test, following the instructions for use. The test will be conducted following both the instructions for the in stream method of sampling and the method of testing when a sample is collected into a container. The results will be compared to those achieved by the study technician.

DETAILED DESCRIPTION:
The study will compare the performance of the Clearblue Advanced Pregnancy Test, when used by consumers according to the instructions for use leaflet (IFUL), and by trained coordinators. Consumer testing will include both sampling in the urine stream and the testing method for urine collected into a container.

In addition, the performance of the Clearblue Advanced Pregnancy Test will be compared to that of the currently marketed Clearblue Digital Pregnancy Test for the detection of pregnancy. In this comparison, both tests will be performed by a trained coordinator using the testing method for urine collected into a container on each volunteer's urine sample.

The study will involve the recruitment of a cross-section of the target pregnancy test users in the United Kingdom, that is, women aged 18-45 who are seeking a pregnancy test. The study will aim to recruit at least 100 volunteers, a minimum of 30 (30%) of whom will be pregnant.

Volunteers will use the Clearblue Advanced Pregnancy Test device using the urine stream method of sampling according to the product instructions. In addition volunteers will be asked to collect a urine sample from the same void and conduct a second Clearblue Advanced Pregnancy Test, using the testing method for urine collected in a container. The volunteer will then complete a study questionnaire on ease of use and leaflet comprehension. The questionnaire, urine sample and used devices will be retained by SPD for evaluation Agreement between the volunteer Pregnancy Test result and study coordinator Pregnancy Test result will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Requiring a pregnancy test
* Willing to provide informed consent and reveal pregnancy status

Exclusion Criteria:

* Employees of SPD. Unipath, Alere or P&G Previous participation in study Previously used Clearblue Advanced Pregnancy Test.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
number of pregnant volunteers as determined by volunteer test result. | 3 months
  Comparison of the performance of the Clearblue Advanced Pregnancy Test in consumer hands when tested using the in-stream method of testing with the performance of the device when used by a study coordinator when testing the same urine sample using the method for urine collected into a container.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline A Parkinson, BSc, Principal Investigator — SPD Development Company Limited
Locations (1):
- SPD Development Company Ltd., Bedford, Bedfordshire, United Kingdom